CLINICAL TRIAL: NCT05279456
Title: A Phase 3b/4 Randomised Trial of 3 Doses of Protein-based Covid-19 Vaccine (SpikoGen)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vaxine Pty Ltd (Industry)
Collaborators: Australian Respiratory and Sleep Medicine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AUST-C19-P3/4
Record Dates: First submitted 2022-03-07; First posted 2022-03-15 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: sars-cov-2; coronavirus; vaccine; adjuvant; Advax; Spikogen; Covax-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — SARS-CoV-2 recombinant spike protein with delta inulin and CpG-ODN adjuvant vaccine

STUDY DESIGN:
Intervention Model Description: Subjects will be stratified for analysis by age, sex and seropositivity at time of study entry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spikogen vaccine - accelerated arm (Experimental): Spikogen vaccine 25 micrograms by intramuscular injection on study months 0, 1 and 2
  Interventions: Biological: Advax-CpG55.2 adjuvanted recombinant spike protein
- Spikogen vaccine - standard arm (Experimental): Spikogen vaccine 25 micrograms by intramuscular injection on study months 0, 1 and 4
  Interventions: Biological: Advax-CpG55.2 adjuvanted recombinant spike protein

INTERVENTIONS:
Biological: Advax-CpG55.2 adjuvanted recombinant spike protein — recombinant SARS-CoV-2 spike protein formulated with Advax-CpG55.2 adjuvant
  Other Names: Spikogen vaccine

SUMMARY:
This study will determine the immunogenicity of Spikogen in vaccine naïve individuals. Spikogen will be administered as two doses 1 month apart with a third booster dose either 1 or 3 months after the second dose. This study will provide key data on SARS-CoV-2 antibody responses.

DETAILED DESCRIPTION:
The SARS-CoV-2 outbreak has caused millions of deaths globally. It has a particularly high mortality rate in elderly people and those with chronic disease where mortality rates can be as high as 20-30%. SARS-COV-2 vaccines remain a key priority to help fight the current pandemic. COVID-19 vaccines prevent symptomatic infection and may help reduce virus transmission. Spikogen® vaccine, also known as Covax-19™ in Australia, is an adjuvanted recombinant protein Covid-19 vaccine has recently been approved by the Iranian FDA for emergency use in Iran in adults as a primary vaccine course and booster dose, after meeting its primary efficacy endpoint in a Phase 3 trial in 16,876 participants randomised 3:1 to receive Spikogen vaccine or saline placebo via two intramuscular doses 3 weeks apart where Spikogen vaccine demonstrated significant protection against serious infection with the delta variant. Approximately 5-10% of the broader Australian population and an even higher proportion of the indigenous populations remains unvaccinated despite current availability of these vaccines. One reason is that some people have medical contraindications to the current vaccines, such as serious allergies to the vaccine components such as polyethyleneglycol (PEG) in the mRNA vaccines.

Spikogen vaccine is made using a recombinant protein approach with the SARS-CoV-2 spike protein synthesized in an insect cell line grown in broth. Insect cell expression of recombinant protein is a well-established vaccine manufacturing approach. Spikogen vaccine also contains a unique Australian developed adjuvant called Advax-CpG55.2, which is added to the spike protein to make the vaccine more effective. AdvaxCpG55.2 has two components, one a natural plant sugar called inulin, and the second a short synthetic oligonucleotide polymer, known as CpG55.2 oligonucleotide.

Spikogen vaccine is designed to protect against SARS-CoV-2 infection. It has been shown to be effective against infection in hamster, ferret and monkey SARS-CoV-2 infection models.

This study will determine the immunogenicity of Spikogen in vaccine-naïve individuals. Spikogen will be administered as two doses 31 month apart with a third booster dose given either 1 or 3 months after the second dose.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Males or females* 18 years of age or older
* Understand and are likely to comply with planned study procedures and be available for all study visits.
* Have not previously had a Covid-19 vaccine and do not intend to have a non-study Covid-19 vaccine within the next 6 months

Exclusion Criteria:

* History of Covid-19 vaccination.
* History of serious vaccine allergy.
* Pregnancy1
* Have received an experimental agent within 30 days prior to the study vaccination or expect to receive another experimental agent during the trial reporting period.
* Any medical, social or mental condition which, in the opinion of the investigator, would be detrimental to the subjects or the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
First dose Seroconversion | 2-4 weeks post first immunisation
  Proportion of subjects in each group stratified by baseline antibody positivity seroconverting to spike protein antibody positivity
Second dose Seroconversion | 2-4 weeks post second immunisation
  Proportion of subjects in each group stratified by baseline antibody positivity seroconverting to spike protein antibody positivity
Third Dose Seroconversion | 2-4 weeks post third immunisation
  Proportion of subjects in each group stratified by baseline antibody positivity seroconverting to spike protein antibody positivity
Final Seroconversion | through study completion, an average of 7 months
  Proportion of subjects in each group stratified by baseline antibody positivity seroconverting to spike protein antibody positivity
First Dose GMT | 2-4 weeks post first immunisation
  Spike protein antibody Geometric Mean Titers (GMT) in each group stratified by baseline antibody positivity
Second Dose GMT | 2-4 weeks post second immunisation
  Spike protein antibody Geometric Mean Titers (GMT) in each group stratified by baseline antibody positivity
Third Dose GMT | 2-4 weeks post third immunisation
  Spike protein antibody Geometric Mean Titers (GMT)in each group stratified by baseline antibody positivity
Final GMT | through study completion, an average of 7 months
  Spike protein antibody Geometric Mean Titers (GMT)in each group stratified by baseline antibody positivity
First Dose Adverse events (AE) | 7 days post first immunisation
  AE occurring within 7 days of immunisation in each group stratified by baseline antibody positivity
Second Dose Adverse events (AE) | 7 days post second immunisation
  AE occurring within 7 days of immunisation in each group stratified by baseline antibody positivity
Third Dose Adverse events (AE) | 7 days post third immunisation
  AE occurring within 7 days of immunisation in each group stratified by baseline antibody positivity
Serious adverse events (SAE) | through study completion, an average of 7 months
  Number of Serious adverse events (SAE) occurring within study period in each group stratified by baseline antibody positivity

SECONDARY OUTCOMES:
First dose Vaccine efficacy | From 2 weeks post-first dose to 2 weeks after second dose
  Proportion of Covid-19 infections in trial participants in each group stratified by baseline antibody positivity
Second dose Vaccine efficacy | From 2 weeks post-second dose to 2 weeks after third dose
  Proportion of Covid-19 infections in trial participants in each group stratified by baseline antibody positivity
Third dose Vaccine efficacy | From 2 weeks post-third dose through study completion, an average of 7 months
  Proportion of Covid-19 infections in trial participants in each group stratified by baseline antibody positivity
Total Covid-19 infections | From first vaccine dose through study completion, an average of 7 months
  Proportion of breakthrough Covid-19 infections in trial participants in each group stratified by baseline antibody positivity
Seroconversion against variants of concern | 2-4 weeks post first, second and third immunisation and at study completion
  Serum spike protein antibody seroconversion rates against each SARS-CoV-2 variant of concern in trial participants in each group stratified by baseline antibody positivity
GMT against variants of concern | 2-4 weeks post first, second and third immunisation and at study completion
  Geometric mean serum spike protein antibodies against SARS-CoV-2 variants in trial participants in each group stratified by baseline antibody positivity

OTHER OUTCOMES:
Antibody kinetics | 2-4 weeks post first, second and third immunisation and at study completion
  rate of change in peak to trough serum spike protein antibody levels over time in each group stratified by baseline antibody positivity
Age effects on seroconversion | 2-4 weeks post first, second and third immunisation and at study completion
  Proprotion seroconverting to spike protein antibodies analysed by age and gender
Age effects on antibody levels | 2-4 weeks post first, second and third immunisation and at study completion
  Geometric Mean Titers of spike protein antibodies in participants by age and gender
immune-deficiency effects on seroconversion | 2-4 weeks post first, second and third immunisation and at study completion
  Proportion of subjects seroconverting to spike protein antibodies in participants with or without immune-deficiency
immune-deficiency effects on antibody levels | 2-4 weeks post first, second and third immunisation and at study completion
  Geometric Mean Titers (GMT) of spike protein antibodies in participants with or without immune-deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Dimitar Sajkov, MBBS, Study Director — ARASMI
Locations (1):
- ARASMI, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share IPD with other researchers, but requests for data access will be considered on a case by case basis

REFERENCES:
- [Background] Li L, Honda-Okubo Y, Huang Y, Jang H, Carlock MA, Baldwin J, Piplani S, Bebin-Blackwell AG, Forgacs D, Sakamoto K, Stella A, Turville S, Chataway T, Colella A, Triccas J, Ross TM, Petrovsky N. Immunisation of ferrets and mice with recombinant SARS-CoV-2 spike protein formulated with Advax-SM adjuvant protects against COVID-19 infection. Vaccine. 2021 Sep 24;39(40):5940-5953. doi: 10.1016/j.vaccine.2021.07.087. Epub 2021 Aug 3. PMID 34420786
- See also: Link to company website — http://vaxine.net